CLINICAL TRIAL: NCT03741153
Title: The Possible Association Between Pseudoexfoliation Syndrome and Diabetes Mellitus in an Egyptian Population
Brief Title: Association Between Pseudoexfoliation Syndrome and Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, gehad salah eldin galal, Principal investigator, Assiut University
Other Study IDs: PXSDM
Record Dates: First submitted 2018-11-11; First posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Lens Diseases
MeSH Terms: conditions — Lens Diseases | interventions — Slit Lamp

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: includes patients who will be diagnosed with Pseudoexfoliation syndrome
  Interventions: Device: slit lamp
- control group: age matched controls who do not have Pseudoexfoliation syndrome
  Interventions: Device: slit lamp

INTERVENTIONS:
Device: slit lamp — 1. Presence of white grayish exfoliation material on the anterior lens capsule and / or the pupillary margin.
  2. Poor pupillary dilatation due to atrophy of the dilator pupillae muscle.
  3. The presence of pseudoexfoliative material (PXF)in cilliary processes and zonules.
  4. presence of PXF material scattered on corneal endothelium.
  5. Flecks of the exfoliative material on the anterior chamber which leads to glaucoma.

SUMMARY:
Pseudoexfoliation syndrome (PEX) is characterized by the deposition of a distinctive fibrillar material in the anterior segment of the eye and was first described in 1917 by Lindberg. It is frequently associated with open angle glaucoma, known as pseudoexfoliation glaucoma, which is one of the most common identifiable forms of secondary open angle glaucoma worldwide. Despite extensive research, the exactchemical nature of the fibrillar material is unknown. It is believed to be secreted multifocally in the iris pigment epithelium, the ciliary epithelium, and the peripheral anterior lens epithelium.

ELIGIBILITY:
Inclusion Criteria:

* Phakic patients presenting to Ophthalmology outpatient clinic Of Assiut University Hospital.

Exclusion Criteria:

* Patients with previous intraocular surgery.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who will be diagnosed with pseudo-exfolian syndrome
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-03-14 (Estimated)

PRIMARY OUTCOMES:
the percentage of diabetic patients with pseudo-exfoliation syndrome | 10 minutes
  slit lamp examination of all diabetic patients to get the percentage of those with pseudo-exfoliation syndrome